CLINICAL TRIAL: NCT03189329
Title: The Effect of Retrobulbar Block on Bi-Hemispheric Cerebral Oxygen Saturation and Early Period Postoperative Cognitive Functions With Lidocaine and Levobupivacaine in Elderly Patients With Ophthalmic Surgery
Brief Title: The Effect of Retrobulbar Block for Eye Surgery on Brain Oxygenation and Cognitive Functions in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cengiz KAYA (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Sponsor-Investigator, Cengiz KAYA, Associate Professor, MD, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PYO.TIP.1904.15.009
Record Dates: First submitted 2017-06-10; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Vitreoretinal Surgery; Cognitive Function Abnormal; Intraoperative Monitoring
Keywords: NIR spectroscopy, cognitive function, eye, nerve block
MeSH Terms: conditions — Cognition Disorders | interventions — Lidocaine; Levobupivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Active Comparator): Patients undergoing block with 2% lidocaine hydrochloride
  Interventions: Drug: 2% lidocaine hydrochloride
- Group LB (Active Comparator): Patients undergoing block with 0.5% levobupivacaine
  Interventions: Drug: 0.5% levobupivacaine

INTERVENTIONS:
Drug: 2% lidocaine hydrochloride — Retrobulbar block was performed with 5 ml of 2% lidocaine hydrochloride (AritmalR, Osel, Istanbul, Turkey) in Group L patients. The block was performed by the same practitioner (fourth year assistant of Ophthalmology Department) using inferotemporal approach as described by Sanderson using 27 gage disposable needles (Atkinson Retrobulbar NeedleR, Asico, USA)
  Arms: Group L
Drug: 0.5% levobupivacaine — and 5ml of 0.5% levobupivacaine (ChirocaineR, Abbvie, Chicago, USA) in Group LB patients. The block was performed by the same practitioner (fourth year assistant of Ophthalmology Department) using inferotemporal approach as described by Sanderson using 27 gage disposable needles (Atkinson Retrobulbar NeedleR, Asico, USA)
  Arms: Group LB

SUMMARY:
The investigators measured changes in cerebral oxygen saturation (rSO2) and MMSE scores after retrobulbar block performed with levobupivacaine and lidocaine in patients undergoing vitreoretinal surgery.A total of 66 patients over the age of 60 undergoing vitreoretinal surgery with a total duration of less than 1 hour were included in this prospective, double-blinded study. The patients were randomly divided into two groups: group L (5ml, 2% lidocaine) and group LB (5ml, 0.5% levobupivacaine). Bilateral rSO2 measurements were recorded before the retrobulbar block and at 1-5 minutes post-block, during the procedure, and at 10-40 minutes post-op. MMSE was performed preoperatively and postoperatively in order to evaluate short term cognitive function. Sensory and motor block durations, pain, akinesia and conjunctival feeling scores, patient-surgeon satisfaction, and complications were also recorded.

DETAILED DESCRIPTION:
A total of 66 patients undergoing vitreoretinal surgery (total duration < 60 minutes) using retrobulbar block, who were classified as category I-III according to the ASA (American Society of Anesthesiologists) Classification system, who were over the age of 60, and who had no cognitive dysfunction were included in the study. Exclusion criteria were as follows: contraindication for retrobulbar block, preoperative systolic blood pressure of 180 mmHg, diastolic blood pressure of above 100 mmHg, uncontrolled diabetes, body mass index ≥ 30 kg/m2, MMSE ≤ 24, advanced organ failure, or Hb < 9gr/dl.The patients were randomly divided into two groups using a sealed-envelope method:

Group L: Patients undergoing block with lidocaine (n = 33) Group LB: Patients undergoing block with levobupivacaine (n = 33) The patients did not undergo premedication in order to accommodate the postoperative MMSE evaluation. For intra-operative sedation, remifentanil (UltivaR, GlaxoSmithKline, Berntford, UK) was initiated as an infusion at a dose range of 0.05-0.1 mcg/kg/min. The mean arterial pressure and heart rate values were allowed to vary up to 20% of the preoperative values of the patients. For this purpose, the remifentanil infusion rate was increased or decreased at the determined dose interval.

Retrobulbar block was performed with 5 ml of 2% lidocaine hydrochloride (AritmalR, Osel, Istanbul, Turkey) in Group L patients and 5ml of 0.5% levobupivacaine (ChirocaineR, Abbvie, Chicago, USA) in Group LB patients. The block was performed by the same practitioner (fourth year assistant of Ophthalmology Department) using inferotemporal approach as described by Sanderson using 27 gage disposable needles (Atkinson Retrobulbar NeedleR, Asico, USA).

Sensory and motor block onset and end times and akinesia score were recorded. The mean arterial pressure (MAP), heart rate (HR), and oxygen saturation (SpO2) were recorded in the preoperative period, at minutes 1, 3, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, and 60 intra-operatively, and at 10, 20, 30, and 40 minutes postoperatively in the recovery room.

. The patients were transferred to the operating table for measurement of bilateral rSO2, and preoxygenation was performed for three minutes using 4 L/min 100% oxygen via nasal cannula. The basal oxygenation values were determined by taking the average of the last 30 s measurements. The rSO2 values were recorded at 1, 3, 5, 10, 15, 20, 25, 30th, 35, 40, 45, 50, 55, and 60 minutes after retrobulbar block, and at 10, 20, 30, and 40 minutes after the completion of the procedure.

Cognitive functions were assessed by the same technician using MMSE in the preoperative period, 40 minutes postoperatively and at 7 days after the operation (short term).Surgeon satisfaction was queried at the end of the case and patient satisfaction was questioned at the end of day.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing vitreoretinal surgery (total duration < 60 minutes)
* The ASA (American Society of Anesthesiologists) Classification I-III
* Over the age of 60
* The patiens who had no cognitive dysfunction

Exclusion Criteria:

* Contraindication for retrobulbar block
* Preoperative systolic blood pressure of 180 mmHg, diastolic blood pressure of above 100 mmHg
* Uncontrolled diabetes
* Body mass index ≥ 30 kg/m2
* MMSE ≤ 24
* Advanced organ failure
* Hb < 9gr/dl

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygen saturation changes (rSO2) | The rSO2 value changes were recorded from baseline up to 40 minutes after surgery
  The NIRS device probes (INVOS-3100AR; Somanetics Inc., Troy, MI, USA) were placed at least 2 cm above the eyebrows and 3 cm away from the mid-line of the forehead, on right and left, in accordance with the instructions of manufacturer.The patient's forehead was cleaned with acetone alcohol before the sensor pads were glued, and wrapped with a bandage so that the sensors were not affected by ambient light. The patients were transferred to the operating table for measurement of bilateral rSO2, and preoxygenation was performed for three minutes using 4 L/min 100% oxygen via nasal cannula.

SECONDARY OUTCOMES:
Cognitive function measurement | Cognitive functions were assessed from baseline up to 7 days after the surgery
  Cognitive functions were assessed by the same technician using the Mini Mental State Examination (MMSE) test.
Sensory block onset time by the conjunctival feeling score using the cotton contact test. | The sensory block onset time was recorded at the beginning of surgery till the first 15 min
  The sensory block onset time was recorded as the moment when the patient did not feel a piece of cotton touching the cornea. This time was measured by the conjunctival feeling score using the cotton contact test (0: normal, 1: less sensitive, 2: complete sensory loss). Score of 2 on the scale was considered as onset time for sensory block.
Sensory block end time by the conjunctival feeling score using the cotton contact test. | The sensory block end time was recorded at the end of surgery till the first 24 h
  The time at which recovery of sensory block was recovered was measured by the conjunctival feeling score using the cotton contact test (0: normal, 1: less sensitive, 2: complete sensory loss). Score of 0 on the scale was considered as end time for sensory block.
Motor block onset time by eye movements score. | The motor block onset time was recorded at the beginning of surgery till the first 15 min
  The motor block onset time was recorded as the time that the patient's eye movements score was four or less. Eye movements score was measured over three points in each of the four quadrants as follows: 3, full eye movement and 0, no movement.
Motor block end time by eye movements score. | The motor block end time was recorded at the end of surgery till the first 24 h
  The time at which recovery of motor block was recovered was measured by the eye movements score (three points in each of the four quadrants as follows: 3, full eye movement and 0, no movement). Score of 12 on the scale was considered as end time for motor block.
The akinesia score measurement | The akinesia score was assessed at the beginning of surgery till the first 15 min.
  The akinesia score was assessed between 0-12 points after 10 minutes of block application. Eye movements were measured over three points in each of the four quadrants as follows: 3, full eye movement and 0, no movement. The sum of the movement scores across all four quadrants was recorded as the akinesian score. An eye with full movement was scored as 12, and an immobile eye was scored as 0. If the akinesia score was four or less, the block was considered successful.
The mean arterial pressure (MAP) measurement | The mean arterial pressure was recorded from baseline up to 40 minutes after surgery
  The mean arterial pressure (MAP) was recorded in the preoperative period, at minutes 1, 3, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, and 60 intra-operatively, and at 10, 20, 30, and 40 minutes postoperatively in the recovery room.
The heart rate (HR) measurement | The heart rate (HR) was recorded from baseline up to 40 minutes after surgery
  The heart rate (HR) was recorded in the preoperative period, at minutes 1, 3, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, and 60 intra-operatively, and at 10, 20, 30, and 40 minutes postoperatively in the recovery room.
The oxygen saturation (SpO2) measurement | The oxygen saturation (SpO2) was recorded from baseline up to 40 minutes after surgery
  The oxygen saturation (SpO2) was recorded in the preoperative period, at minutes 1, 3, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, and 60 intra-operatively, and at 10, 20, 30, and 40 minutes postoperatively in the recovery room.
Surgeon satisfaction | Surgeon satisfaction was queried at the end of the surgery till the first 15 min.
  They were asked to score over 10 point scale. Surgeon satisfaction was evaluated using 10 point scale ( 0 = not satisfied at all and 10 = very satisfied)
Patient satisfaction | Patient satisfaction was questioned 24 hours after surgery
  They were asked to score over 10 point scale. Patient satisfaction was evaluated using 10 point scale ( 0 = not satisfied at all and 10 = very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Cengiz Kaya, MD, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis Universitesi, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen RC, Doody R, Kurz A, Mohs RC, Morris JC, Rabins PV, Ritchie K, Rossor M, Thal L, Winblad B. Current concepts in mild cognitive impairment. Arch Neurol. 2001 Dec;58(12):1985-92. doi: 10.1001/archneur.58.12.1985. PMID 11735772
- [Background] Ripart J, Lefrant JY, Vivien B, Charavel P, Fabbro-Peray P, Jaussaud A, Dupeyron G, Eledjam JJ. Ophthalmic regional anesthesia: medial canthus episcleral (sub-tenon) anesthesia is more efficient than peribulbar anesthesia: A double-blind randomized study. Anesthesiology. 2000 May;92(5):1278-85. doi: 10.1097/00000542-200005000-00015. PMID 10781272
- [Background] BOBERG-ANS J. Experience in clinical examination of corneal sensitivity; corneal sensitivity and the naso-lacrimal reflex after retrobulbar anaesthesia. Br J Ophthalmol. 1955 Dec;39(12):705-26. doi: 10.1136/bjo.39.12.705. No abstract available. PMID 13276583
- [Background] Wang PW, Chen ML, Huang LW, Yang W, Wu KY, Huang YF. Prenatal nonylphenol exposure, oxidative and nitrative stress, and birth outcomes: A cohort study in Taiwan. Environ Pollut. 2015 Dec;207:145-51. doi: 10.1016/j.envpol.2015.08.044. Epub 2015 Sep 12. PMID 26367708
- [Background] Tsai TC, Orav EJ, Jha AK. Patient satisfaction and quality of surgical care in US hospitals. Ann Surg. 2015 Jan;261(1):2-8. doi: 10.1097/SLA.0000000000000765. PMID 24887985
- [Background] Casati A, Fanelli G, Pietropaoli P, Proietti R, Tufano R, Montanini S; Collaborative Italian Study Group on Anaesthesia in Elderly Patients; Danelli G, Nuzzi M, Mentegazzi F, Torri G, Martani C, Spreafico E, Fierro G, Pugliese F, De Cosmo G, Aceto P, Servillo G, Monaco F. Monitoring cerebral oxygen saturation in elderly patients undergoing general abdominal surgery: a prospective cohort study. Eur J Anaesthesiol. 2007 Jan;24(1):59-65. doi: 10.1017/S0265021506001025. Epub 2006 Jul 7. PMID 16824246
- [Result] Astrup J. Energy-requiring cell functions in the ischemic brain. Their critical supply and possible inhibition in protective therapy. J Neurosurg. 1982 Apr;56(4):482-97. doi: 10.3171/jns.1982.56.4.0482. No abstract available. PMID 6278105
- [Result] Shokunbi MT, Gelb AW, Wu XM, Miller DJ. Continuous lidocaine infusion and focal feline cerebral ischemia. Stroke. 1990 Jan;21(1):107-11. doi: 10.1161/01.str.21.1.107. PMID 2300976
- [Result] Rasool N, Faroqui M, Rubinstein EH. Lidocaine accelerates neuroelectrical recovery after incomplete global ischemia in rabbits. Stroke. 1990 Jun;21(6):929-35. doi: 10.1161/01.str.21.6.929. PMID 2349597
- [Result] Haschke RH, Fink BR. Lidocaine effects on brain mitochondrial metabolism in vitro. Anesthesiology. 1975 Jun;42(6):737-40. doi: 10.1097/00000542-197506000-00018. PMID 1130742
- [Result] Baik JS, Sohn JT, Ok SH, Kim JG, Sung HJ, Park SS, Park JY, Hwang EM, Chung YK. Levobupivacaine-induced contraction of isolated rat aorta is calcium dependent. Can J Physiol Pharmacol. 2011 Jul;89(7):467-76. doi: 10.1139/y11-046. Epub 2011 Jul 21. PMID 21812525
- [Result] Sung HJ, Ok SH, Sohn JY, Son YH, Kim JK, Lee SH, Han JY, Lim DH, Shin IW, Lee HK, Chung YK, Choi MJ, Sohn JT. Vasoconstriction potency induced by aminoamide local anesthetics correlates with lipid solubility. J Biomed Biotechnol. 2012;2012:170958. doi: 10.1155/2012/170958. Epub 2012 Jun 17. PMID 22778542
- [Result] Birt DJ, Cummings GC. The efficacy and safety of 0.75% levobupivacaine vs 0.75% bupivacaine for peribulbar anaesthesia. Eye (Lond). 2003 Mar;17(2):200-6. doi: 10.1038/sj.eye.6700313. PMID 12640407
- [Result] Suehiro K, Okutai R. Duration of cerebral desaturation time during single-lung ventilation correlates with mini mental state examination score. J Anesth. 2011 Jun;25(3):345-9. doi: 10.1007/s00540-011-1136-1. Epub 2011 Apr 12. PMID 21484501
- [Result] Zhang Y, Qian Y, Bao H, Shi H, Zhou J. [Effect of Stellate Ganglion Block on Bilateral Regional Cerebral Oxygen Saturation and Postoperative Cognitive Function]. Sheng Wu Yi Xue Gong Cheng Xue Za Zhi. 2016 Feb;33(1):132-5. Chinese. PMID 27382753
- [Result] Aksu R, Bicer C, Ozkiris A, Akin A, Bayram A, Boyaci A. Comparison of 0.5% levobupivacaine, 0.5% bupivacaine, and 2% lidocaine for retrobulbar anesthesia in vitreoretinal surgery. Eur J Ophthalmol. 2009 Mar-Apr;19(2):280-4. doi: 10.1177/112067210901900217. PMID 19253247
- [Result] Simonson D. Retrobulbar block: a review for the clinician. AANA J. 1990 Dec;58(6):456-61. PMID 2102683
- [Result] Murphy PJ, Lawrenson JG, Patel S, Marshall J. Reliability of the non-contact corneal aesthesiometer and its comparison with the Cochet-Bonnet aesthesiometer. Ophthalmic Physiol Opt. 1998 Nov;18(6):532-9. PMID 10070549
- [Result] Pacella E, Collini S, Pacella F, Piraino DC, Santamaria V, De Blasi RA. Levobupivacaine vs. racemic bupivacaine in peribulbar anaesthesia: a randomized double blind study in ophthalmic surgery. Eur Rev Med Pharmacol Sci. 2010 Jun;14(6):539-44. PMID 20712261
- [Result] Ghali AM. The efficacy of 0.75% levobupivacaine versus 0.75% ropivacaine for peribulbar anesthesia in vitreoretinal surgery. Saudi J Anaesth. 2012 Jan;6(1):22-6. doi: 10.4103/1658-354X.93050. PMID 22412772
- [Result] Kim MN, Durduran T, Frangos S, Edlow BL, Buckley EM, Moss HE, Zhou C, Yu G, Choe R, Maloney-Wilensky E, Wolf RL, Grady MS, Greenberg JH, Levine JM, Yodh AG, Detre JA, Kofke WA. Noninvasive measurement of cerebral blood flow and blood oxygenation using near-infrared and diffuse correlation spectroscopies in critically brain-injured adults. Neurocrit Care. 2010 Apr;12(2):173-80. doi: 10.1007/s12028-009-9305-x. PMID 19908166